CLINICAL TRIAL: NCT04519801
Title: Blood Flow Restriction Therapy for the Post-Operative Rehabilitation of Anterior Cruciate Ligament Reconstruction With Quadriceps Tendon Autograft: A Randomized, Controlled Trial
Brief Title: BFR Therapy for Post-Op Rehab of ACL Reconstruction With Quadriceps Tendon Autograft
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: American Orthopaedic Society for Sports Medicine (Other); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Daniel Cognetti, Director of Clinical Research, Principal Investigator, Staff Orthopaedic Surgeon, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C.2020.053
Record Dates: First submitted 2020-08-14; First posted 2020-08-20 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: ACL Injury
Keywords: BFR; ACLR; Quadriceps Tendon
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either REHAB or REHAB + BFR (study intervention) using a block randomization scheme.
Who Masked: Investigator
Masking Description: The operating surgeon will remain blinded to the post-operative rehabilitation regimen to which subjects are randomized to post-operative rehabilitation regimen (REHAB vs. REHAB + BFR.)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- REHAB (Other): Standard post-operative rehabilitation regimen (REHAB) (Control)
  Interventions: Other: Standard REHAB
- REHAB + BFR (Experimental): Standard rehabilitation regimen with BFR therapy (REHAB + BFR) (Experimental)
  Interventions: Other: Blood Flow Restriction (BFR) therapy; Other: Standard REHAB

INTERVENTIONS:
Other: Blood Flow Restriction (BFR) therapy — BFR therapy beginning after first MD follow up appointment after ACL reconstruction with quadriceps tendon autograft and the following functional criteria have been met: 1.) incisions healing or healed without signs of infection or dehiscence. 2.) ROM to at least 90 degree flexion. 3.) Able to perform unilateral weight bearing for 5 seconds. 4.) Pain under control and minimal knee effusion.
  Arms: REHAB + BFR
Other: Standard REHAB — Standard post-operative rehabilitation regimen (REHAB) beginning after first MD follow up appointment ACL reconstruction with quadriceps tendon autograft and the following functional criteria have been met: 1.) incisions healing or healed without signs of infection or dehiscence. 2.) ROM to at least 90 degree flexion. 3.) Able to perform unilateral weight bearing for 5 seconds. 4.) Pain under control and minimal knee effusion

SUMMARY:
The overall objective of the proposed research is to conduct a prospective, randomized controlled trial to investigate whether the addition of BFR therapy to standard post-operative rehabilitation regimen significantly improves clinical outcomes following anterior cruciate ligament reconstruction (ACLR) standardized with respect to both surgical technique and graft selection. Patients indicated for ACLR will be screened and offered enrollment into this prospective, randomized controlled trial. MRI of bilateral thighs will be performed within 7 days of ACLR. Patients will be randomized to either REHAB or REHAB + BFR (study intervention) using a block randomization scheme. Patients will undergo repeat MRI of bilateral thighs pre-surgery, at 12 weeks, and at 52 weeks post-operatively (primary outcome measure.) Patient reported outcome (PRO) instruments will be administered pre-operatively to establish pre-operative debility related to ACL injury and subsequently after ACLR at 24 weeks, 36 weeks, and 52 weeks post-operative (secondary outcome measures).

DETAILED DESCRIPTION:
The overall objective of the proposed research is to conduct a prospective, randomized controlled trial to investigate whether the addition of BFR therapy to standard post-operative rehabilitation regimen significantly improves clinical outcomes following ACLR standardized with respect to both surgical technique and graft selection. The investigator's central hypothesis is that the addition of BFR therapy has the potential to accelerate surgical recovery, expedite return-to-duty, and maximize medical readiness following ACLR. In the proposed trial validated patient reported outcome measures will be used to assess for functional clinical improvement, while quadriceps musculature cross sectional area (CSA) as measured on MRI will be used to quantify the effect of therapy on quadriceps strength. The rationale for using this modality is based upon the fact that the measurement of quadriceps CSA and muscle volume as surrogates for overall quadriceps function is well described, and a number of studies have convincingly demonstrated positive correlations between these parameters and quadriceps strength4, 17. However, in spite of these reports, the acceptance acknowledging MRI as a surrogate for quadriceps strength remains limited. Therefore, isokinetic and isometric quadriceps strength of both the operative and non-operative knee extensors (quadriceps) will be measured pre-operatively within 7-10 days approximately prior to ACLR and post-operatively at approximately 12 weeks, 24 weeks, 36 weeks, and 52 weeks. MRI of bilateral thighs will be performed immediately prior to ACLR to establish a baseline CSA in the operative and non-operative lower extremity. Then a repeat MRI will be performed following the conclusion of a standardized 12-week (approximately) post-operative rehabilitation regimen among patients randomized to either a standard rehabilitation regimen (REHAB) or a rehabilitation regimen with BFR (REHAB + BFR.) Finally, MRI will be repeated at 52 weeks post-operative to examine for latent changes in CSA once patients have been returned to unrestricted physical activities.

AIM 1: To determine if the addition of BFR therapy to a standard post-operative rehabilitation protocol increases quadriceps muscle cross sectional area and volume after ACLR as measured with magnetic resonance imaging (MRI).

Hypothesis: The addition of BFR therapy to a standard post-operative rehabilitation regimen following ACLR will increase quadriceps muscle CSA and volume when compared to a standard post-operative rehabilitation regimen measured at approximately 12-weeks post-operative.

AIM 2: To determine if any observed increases in quadriceps muscle CSA and volume are sustained beyond the cessation of BFR therapy at approximately 12-weeks post-operative by performing repeat MRI at 52 weeks post-operative.

Hypothesis: Observed increases in quadriceps muscle CSA and volume will be sustained beyond the cessation of BFR therapy at 52 weeks post-operative.

AIM 3: To determine if CSA measurements obtained by MRI reliably predict knee extensor strength.

Hypothesis: CSA measurements obtained by MRI reliably predict knee extensor strength as measured by isokinetic and isometric testing.

AIM 4: To determine if the addition of BFR therapy to a standard post-operative rehabilitation regimen following ACLR results in significantly improved functional outcomes when compared to a standard post-operative rehabilitation regimen at 24, 36, and 52 weeks post-operative using patient reported outcomes (PRO).

Hypothesis: The addition of BFR therapy to a standard post-operative rehabilitation regimen following ACLR will result in significantly improved PRO when compared to a standard post-operative rehabilitation regimen at 24, 36, and 52-weeks post-operative.

ELIGIBILITY:
Inclusion Criteria:

* Active duty member or Department of Defense Military Health System beneficiary
* 15 to 45 years of age
* Indicated for ACL reconstruction with quadriceps tendon autograft with evidence of skeletal maturity; no open physes/growth plates

Exclusion Criteria:

* Patients undergoing a concomitant surgical procedure that would otherwise require a period of immobilization and/or restricted weight bearing (i.e. meniscal repair, meniscal allograft transplantation, osteochondral allograft transplantation, high tibial osteotomy) will be excluded.
* Undergoing combined multiligamentous knee injury reconstruction
* Unable to consistently participate in the prescribed post-operative rehabilitation regimen
* No patients with a history of recent lower extremity deep vein thrombosis, within the 12 months or on active treatment with anticoagulants, a history of ipsilateral lower extremity lymph node dissection or a history of endothelial dysfunction.
* Patients that are unable to obtain MRI secondary to either intolerance and/or implanted medical devices that preclude the safe completion of the MRI.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Quadriceps CSA MRI | [Timeframe: within 7-10 days of ACLR] [Time Frame: approximately 12-14 weeks post operative] [Time Frame: approximately 52-54 weeks post-operative]
  Quadriceps CSA as measured on MRI
Knee extensor strength | [Time Frame: approximately withing 7-10 days of ACLR] [Time Frame: 12 weeks post operatively] [Time Frame: 24 weeks post-operatively] [Time Frame: 36 weeks post-operatively] [Time Frame: 52 weeks post-operatively]
  Knee extensor isokinetic and isometric strength measurements

SECONDARY OUTCOMES:
Patient Reported Outcome - Pain on 10 cm Visual Analog Scale (VAS) | [Time Frame: pre-operatively] [Time Frame: 6 months post-operatively] [Time Frame: 9 months post-operatively] [Time Frame: 12 months post-operatively]
  The VAS is a unidimensional measure of pain intensity that has been frequently reported among adults. The simplest VAS is represented as a horizontal 10 cm line. The ends are defined as the extreme limits of parameter being measured (e.g. pain) oriented from the left (worst) to the right (best.) Patients are asked mark their perceived level of pain on the horizontal line. The VAS score is determined by measuring in mm from the left hand end of the horizontal line to where the patient marks. A higher score represents greater pain intensity.
Patient Reported Outcome - Lyscholms Score | [Time Frame: pre-operatively] [Time Frame: 6 months post-operatively] [Time Frame: 9 months post-operatively] [Time Frame: 12 months post-operatively]
  Comprised of 8 items (limp, support, locking, instability, pain, swelling, stair climbing, squatting), which patients are asked a series of questions to characterize their experiences with respect to each of these 8 items. Patients' responses are summed, with a score of 100 denoting no symptoms or debility.
Patient Reported Outcome - International Knee Documentation Committee Form (IKDC) | [Time Frame: pre-operatively] [Time Frame: 6 months post-operatively] [Time Frame: 9 months post-operatively] [Time Frame: 12 months post-operatively]
  This questionnaire is broken down into three categories: symptoms, sports activity, and knee function. The symptoms subscale focuses on an assessment of pain, stiffness, swelling, and the sensation of "giving-way" of the knee. The sports activity subscale focuses on completion of tasks such as going up and down stairs, rising from a seated position, squatting, and jumping. The knee function subscale asks the respondent to characterize their knee at present versus prior to injury. The IKDC is scored out of 100 points, with a score of 100 representing optimal knee function.
Patient Reported Outcome - Knee Osteoarthritis Outcome Score (KOOS) | [Time Frame: pre-operatively] [Time Frame: 6 months post-operatively] [Time Frame: 9 months post-operatively] [Time Frame: 12 months post-operatively]
  The KOOS is a comprehensive scoring system that evaluates both short and long-term consequence of knee injury. It is comprised of 42 items, which are scored separately in 5 subscales (pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and knee-related quality of life (5 items).) Among the strengths of the KOOS as a PRO is its inclusion of two different subscales for physical function relating to daily life, sport, and recreation. A score of 100 represents no knee symptoms, which is then converted to a percentage score to characterize a patient's overall satisfaction with their knee function.
Connor-Davidson Resilience Scale (CD-RISC) | [Time Frame: pre-operatively] [Time Frame: 6 months post-operatively] [Time Frame: 9 months post-operatively] [Time Frame: 12 months post-operatively]
  The CD- RISC 2, 10, or 25 item validated instrument that is self-rated assessment of psychological resiliency. This instrument has shown reliability in measuring the ability to adapt to change, the ability to deal with what comes along, the ability to cope with stress, the ability to stay focused and think clearly, the ability to not get discouraged in the face of failure, the ability to handle unpleasant feelings such as anger, pain or sadness.
Anterior Cruciate Ligament Return to Sport after Injury (ACL-RSI) (Short version 6Q) | [Time Frame: pre-operatively] [Time Frame: 6 months post-operatively] [Time Frame: 9 months post-operatively] [Time Frame: 12 months post-operatively]
  ACL-RSI instrument measure one's emotion, confidence, and risk appraisal when returning to sports after an ACL injury and/or reconstructive surgery. The survey consists of 12 items that are graded on a visual analogue scale from 0 points (extremely negative psychological responses) to 100 points (no negative psychological responses). The results of the survey have been found to be strongly and significantly associated with return to sport.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Sheean, MD, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center- Clinical Research Center, San Antonio, Texas, United States

REFERENCES:
- [Background] Sanders TL, Maradit Kremers H, Bryan AJ, Larson DR, Dahm DL, Levy BA, Stuart MJ, Krych AJ. Incidence of Anterior Cruciate Ligament Tears and Reconstruction: A 21-Year Population-Based Study. Am J Sports Med. 2016 Jun;44(6):1502-7. doi: 10.1177/0363546516629944. Epub 2016 Feb 26. PMID 26920430
- [Background] Goetschius J, Hart JM. Knee-Extension Torque Variability and Subjective Knee Function in Patients with a History of Anterior Cruciate Ligament Reconstruction. J Athl Train. 2016 Jan;51(1):22-7. doi: 10.4085/1062-6050-51.1.12. Epub 2015 Dec 31. PMID 26720104
- [Background] Zwolski C, Schmitt LC, Quatman-Yates C, Thomas S, Hewett TE, Paterno MV. The influence of quadriceps strength asymmetry on patient-reported function at time of return to sport after anterior cruciate ligament reconstruction. Am J Sports Med. 2015 Sep;43(9):2242-9. doi: 10.1177/0363546515591258. Epub 2015 Jul 16. PMID 26183172
- [Background] Thomas AC, Wojtys EM, Brandon C, Palmieri-Smith RM. Muscle atrophy contributes to quadriceps weakness after anterior cruciate ligament reconstruction. J Sci Med Sport. 2016 Jan;19(1):7-11. doi: 10.1016/j.jsams.2014.12.009. Epub 2015 Jan 13. PMID 25683732
- [Background] Kuenze C, Hertel J, Saliba S, Diduch DR, Weltman A, Hart JM. Clinical thresholds for quadriceps assessment after anterior cruciate ligament reconstruction. J Sport Rehabil. 2015 Feb;24(1):36-46. doi: 10.1123/jsr.2013-0110. Epub 2014 Sep 8. PMID 25203517
- [Background] Johnston PT, McClelland JA, Webster KE. Lower Limb Biomechanics During Single-Leg Landings Following Anterior Cruciate Ligament Reconstruction: A Systematic Review and Meta-Analysis. Sports Med. 2018 Sep;48(9):2103-2126. doi: 10.1007/s40279-018-0942-0. PMID 29949109
- [Background] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Background] Burgomaster KA, Moore DR, Schofield LM, Phillips SM, Sale DG, Gibala MJ. Resistance training with vascular occlusion: metabolic adaptations in human muscle. Med Sci Sports Exerc. 2003 Jul;35(7):1203-8. doi: 10.1249/01.MSS.0000074458.71025.71. PMID 12840643
- [Background] Takarada Y, Tsuruta T, Ishii N. Cooperative effects of exercise and occlusive stimuli on muscular function in low-intensity resistance exercise with moderate vascular occlusion. Jpn J Physiol. 2004 Dec;54(6):585-92. doi: 10.2170/jjphysiol.54.585. PMID 15760491
- [Background] Loenneke JP, Kim D, Fahs CA, Thiebaud RS, Abe T, Larson RD, Bemben DA, Bemben MG. Effects of exercise with and without different degrees of blood flow restriction on torque and muscle activation. Muscle Nerve. 2015 May;51(5):713-21. doi: 10.1002/mus.24448. PMID 25187395
- [Background] Hughes L, Paton B, Rosenblatt B, Gissane C, Patterson SD. Blood flow restriction training in clinical musculoskeletal rehabilitation: a systematic review and meta-analysis. Br J Sports Med. 2017 Jul;51(13):1003-1011. doi: 10.1136/bjsports-2016-097071. Epub 2017 Mar 4. PMID 28259850
- [Background] Loenneke JP, Wilson JM, Wilson GJ, Pujol TJ, Bemben MG. Potential safety issues with blood flow restriction training. Scand J Med Sci Sports. 2011 Aug;21(4):510-8. doi: 10.1111/j.1600-0838.2010.01290.x. Epub 2011 Mar 16. PMID 21410544
- [Background] DePhillipo NN, Kennedy MI, Aman ZS, Bernhardson AS, O'Brien L, LaPrade RF. Blood Flow Restriction Therapy After Knee Surgery: Indications, Safety Considerations, and Postoperative Protocol. Arthrosc Tech. 2018 Sep 24;7(10):e1037-e1043. doi: 10.1016/j.eats.2018.06.010. eCollection 2018 Oct. PMID 30377584
- [Background] Tennent DJ, Hylden CM, Johnson AE, Burns TC, Wilken JM, Owens JG. Blood Flow Restriction Training After Knee Arthroscopy: A Randomized Controlled Pilot Study. Clin J Sport Med. 2017 May;27(3):245-252. doi: 10.1097/JSM.0000000000000377. PMID 27749358
- [Background] Iversen E, Rostad V, Larmo A. Intermittent blood flow restriction does not reduce atrophy following anterior cruciate ligament reconstruction. J Sport Health Sci. 2016 Mar;5(1):115-118. doi: 10.1016/j.jshs.2014.12.005. Epub 2015 Apr 18. PMID 30356481
- [Background] Takarada Y, Takazawa H, Ishii N. Applications of vascular occlusion diminish disuse atrophy of knee extensor muscles. Med Sci Sports Exerc. 2000 Dec;32(12):2035-9. doi: 10.1097/00005768-200012000-00011. PMID 11128848
- [Background] Kuenze CM, Blemker SS, Hart JM. Quadriceps function relates to muscle size following ACL reconstruction. J Orthop Res. 2016 Sep;34(9):1656-62. doi: 10.1002/jor.23166. Epub 2016 Jan 27. PMID 26763833
- [Background] Sheean AJ, Musahl V, Slone HS, Xerogeanes JW, Milinkovic D, Fink C, Hoser C; International Quadriceps Tendon Interest Group. Quadriceps tendon autograft for arthroscopic knee ligament reconstruction: use it now, use it often. Br J Sports Med. 2018 Jun;52(11):698-701. doi: 10.1136/bjsports-2017-098769. Epub 2018 Apr 28. PMID 29705749
- [Background] Samuelsen BT, Webster KE, Johnson NR, Hewett TE, Krych AJ. Hamstring Autograft versus Patellar Tendon Autograft for ACL Reconstruction: Is There a Difference in Graft Failure Rate? A Meta-analysis of 47,613 Patients. Clin Orthop Relat Res. 2017 Oct;475(10):2459-2468. doi: 10.1007/s11999-017-5278-9. PMID 28205075
- [Background] Myles PS, Myles DB, Galagher W, Boyd D, Chew C, MacDonald N, Dennis A. Measuring acute postoperative pain using the visual analog scale: the minimal clinically important difference and patient acceptable symptom state. Br J Anaesth. 2017 Mar 1;118(3):424-429. doi: 10.1093/bja/aew466. PMID 28186223
- [Background] Briggs KK, Steadman JR, Hay CJ, Hines SL. Lysholm score and Tegner activity level in individuals with normal knees. Am J Sports Med. 2009 May;37(5):898-901. doi: 10.1177/0363546508330149. Epub 2009 Mar 23. PMID 19307332
- [Background] Ra HJ, Kim HS, Choi JY, Ha JK, Kim JY, Kim JG. Comparison of the ceiling effect in the Lysholm score and the IKDC subjective score for assessing functional outcome after ACL reconstruction. Knee. 2014 Oct;21(5):906-10. doi: 10.1016/j.knee.2014.06.004. Epub 2014 Jun 21. PMID 24998912
- [Background] Grevnerts HT, Terwee CB, Kvist J. The measurement properties of the IKDC-subjective knee form. Knee Surg Sports Traumatol Arthrosc. 2015 Dec;23(12):3698-706. doi: 10.1007/s00167-014-3283-z. Epub 2014 Sep 6. PMID 25193574
- [Background] Gerber JP, Marcus RL, Dibble LE, Greis PE, Burks RT, LaStayo PC. Effects of early progressive eccentric exercise on muscle structure after anterior cruciate ligament reconstruction. J Bone Joint Surg Am. 2007 Mar;89(3):559-70. doi: 10.2106/JBJS.F.00385. PMID 17332105
- [Background] Agarwalla A, Puzzitiello RN, Liu JN, Cvetanovich GL, Gowd AK, Verma NN, Cole BJ, Forsythe B. Timeline for Maximal Subjective Outcome Improvement After Anterior Cruciate Ligament Reconstruction. Am J Sports Med. 2019 Aug;47(10):2501-2509. doi: 10.1177/0363546518803365. Epub 2018 Nov 12. PMID 30419175
- [Background] Prue J, Roman DP, Giampetruzzi NG, Fredericks A, Lolic A, Crepeau A, Pace JL, Weaver AP. Side Effects and Patient Tolerance with the Use of Blood Flow Restriction Training after ACL Reconstruction in Adolescents: A Pilot Study. Int J Sports Phys Ther. 2022 Apr 2;17(3):347-354. doi: 10.26603/001c.32479. eCollection 2022. PMID 35391873